CLINICAL TRIAL: NCT00427167
Title: Phase I Study of the Safety and Immunogenicity of AMA1-C1/Alhydrogel + CPG 7909, an Asexual Blood Stage Vaccine for Plasmodium Falciparum Malaria
Brief Title: Phase I Study of AMA1-C1/Alhydrogel® (Registered Trademark) + CPG 7909 Malaria Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 070083; 07-I-0083
Record Dates: First submitted 2007-01-25; First posted 2007-01-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-08-03

CONDITIONS: Malaria
Keywords: Blood Stage; Investigational; Vaccine; Malaria; Healthy Volunteer; HV
MeSH Terms: conditions — Malaria | interventions — ProMune; Sodium Chloride; Phosphates

INTERVENTIONS:
Biological: AMA1-C1/Alhydrogel + CPG 7909 (Saline)
Biological: AMA1-C1/Alhydrogel + CPG 7909 (Phosphate)
Drug: AMA1-C1/Alhydrogel + CPG 7909

SUMMARY:
This study will evaluate the safety and immune response of healthy volunteers to an experimental malaria vaccine called AMA1-C1/Alhydrogel® (Registered Trademark) + CPG 7909. Malaria is an infection of red blood cells caused by a parasite, Plasmodium falciparum, that is spread by certain kinds of mosquitoes. Each year, about 1 million people are killed by malaria worldwide, most of them young children in Africa. AMA1 C1 may help block the malaria parasite from getting into red blood cells. The vaccine is mixed with Alhydrogel® (Registered Trademark), a material that is commonly added to vaccines to make them work better (also called an adjuvant). Besides evaluating the vaccine, this study will also test two solutions of an experimental adjuvant, CPG 7909-P and CPG 7909-S.

Healthy people between 18 and 50 years of age may be eligible for this 7-month study. Participants are randomly assigned to one of four treatment groups (A, B, C or D below). All receive two vaccinations, given as a shot in the upper arm either 1 or 2 months apart, as shown:

* Group A: AMA1 CI/Alhydrogel® (Registered Trademark)/CPG 7909-P at Day 0 and Day 28 (1-month interval)
* Group B: AMA1 CI/Alhydrogel® (Registered Trademark)/CPG 7909-S at Day 0 and Day 28 (1-month interval)
* Group C: AMA1 CI/Alhydrogel® (Registered Trademark)/CPG 7909-P at Day 0 and Day 56 (2-month interval)
* Group D: AMA1 CI/Alhydrogel® (Registered Trademark)/CPG 7909-S at Day 0 and Day 56 (2-month interval)

Group A and B participants return to the clinic for checkups at 3, 7, and 14 days after each vaccination and again at months 2, 3, 4, 5, and 7. Group C and D participants come to the clinic at 3, 7, and 14 days after each vaccination and again at months 3, 4, 5, and 7.

In addition to the vaccinations, the study includes the following procedures:

* Photographs of the subject's arm where the vaccination is given if a rash develops.
* Daily temperature and symptoms record for the first 6 days after each of the 2 vaccinations, and at any other time there is concern about fever or other symptoms.
* Blood draws about 12 times during the study to check for safety and to measure the antibody response and the effect of the study vaccine.

Some participants may be asked to undergo plasmapheresis, a procedure for collecting plasma, the liquid part of the blood. This is done by using a machine called a blood cell separator. Blood is collected through a needle place...

DETAILED DESCRIPTION:
AMA1-C1 + CPG 7909 is a blood stage malaria vaccine candidate. The objectives of this Phase 1 study are to confirm the previously demonstrated safety and immunogenicity of AMA1-C1 + CPG 7909 formulated in a phosphate buffer. In addition, this study will evaluate the safety and immunogenicity of AMA1-C1 + CPG 7909 formulated in a saline buffer, and determine if the addition of CPG 7909 in a saline buffer enhances the immune response to AMA1-C1 in a manner similar to that seen with the addition of CPG 7909 in a phosphate buffer. The immunological effect of giving a second dose of vaccine at 1 or 2 months will also be evaluated. The study is a double blind Phase 1 clinical trial in healthy adult volunteers. Volunteers will be screened and 24 participants will be enrolled and randomly assigned to 1 of 4 groups in a 2x2 design: 6 volunteers will receive 2 doses of 80 micrograms AMA1-C1/Alhydrogel + 500 micrograms CPG 7909 (phosphate) at a 1-month dosing interval; 6 volunteers will receive 2 doses of 80 micrograms AMA1-C1/Alhydrogel + 500 micrograms CPG 7909 (saline) at a 1 month dosing interval; 6 volunteers will receive 2 doses of 80 micrograms AMA1-C1/Alhydrogel + 500 micrograms CPG 7909 (phosphate) at a 2-month dosing interval; and 6 volunteers will receive 2 doses of 80 micrograms AMA1-C1/Alhydrogel + 500 micrograms CPG 7909 (saline) at a 2 month dosing interval. Safety outcome measures are local and systemic (including laboratory) adverse events. Immune responses to vaccination will be measured by enzyme-linked immunosorbent assay (ELISA) and parasite growth inhibition assay (GIA), and will be compared among groups.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age between 18 and 50 years, inclusive.

Good general health as determined by review of medical history and/or clinical tests at screening.

Available for the duration of the trial (30 weeks).

Willingness to participate in the study as evidenced by signing the informed consent document.

EXCLUSION CRITERIA:

1. Pregnancy as determined by a positive urine beta-hCG at any time during the study (if female).
2. Participant unwilling to use reliable contraception methods for at least 2 weeks prior to vaccination and for the duration of the trial. Reliable methods of birth control include: pharmacologic contraceptives including oral, parenteral, and transcutaneous delivery; condoms with spermicide; diaphragm with spermicide; surgical sterilization; vaginal ring; intrauterine device; abstinence; and post-menopause (if female).
3. Currently breast-feeding (if female).
4. Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the study protocol.
5. Neutropenia as defined by an absolute neutrophil count less than 1500/mm(3).
6. Alanine aminotransaminase (ALT) level above the laboratory-defined upper limit of normal.
7. Serum creatinine level above the laboratory-defined upper limit of normal.
8. Hemoglobin below the laboratory-defined lower limit of normal, by sex.
9. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies including urinalysis.
10. Other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant participating in the trial or would render the subject unable to comply with the protocol.
11. History of receiving any investigational product within the past 30 days.
12. Participant has had medical, occupational or family problems as a result of alcohol or illicit drug use during the past 12 months.
13. History of a severe allergic reaction or anaphylaxis.
14. Positive ELISA and confirmatory Western blot tests for HIV-1.
15. Positive ELISA and confirmatory immunoblot tests for hepatitis C virus (HCV).
16. Positive hepatitis B surface antigen (HBsAg) by ELISA.
17. Pre-existing autoimmune or antibody-mediated diseases including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, or autoimmune thrombocytopenia.
18. Known immunodeficiency syndrome.
19. Positive serum anti-dsDNA titer.
20. Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days of starting this study.
21. Receipt of a live vaccine within past 4 weeks or a killed vaccine within past 2 weeks prior to entry into the study.
22. History of a surgical splenectomy.
23. Receipt of blood products within the past 6 months.
24. Previous receipt of an investigational malaria vaccine.
25. Receipt of antimalarial prophylaxis during the past 12 months, or receipt of chloroquine or related compounds (amodiaquine or primaquine) in the previous 8 weeks prior to study entry.
26. Prior malaria infection.
27. Any medical, psychiatric, social, or occupational condition or other responsibility that, in the judgment of the Principal Investigator (PI), would interfere with the evaluation of study objectives.
28. History of a known allergy to nickel.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300
Dates: Start 2007-01-23; Primary Completion 2008-11-05 (Actual); Study Completion 2008-11-05 (Actual)

PRIMARY OUTCOMES:
Assessment of the safety and reactogenicity of the AMA1-C1/Alhydrogel + CPG 7909 vaccine in phosphate and saline buffers; and determine the frequency of summarized systemic and local AFs by severity and relationship to the vaccine.

SECONDARY OUTCOMES:
Demonstrate that the immune responses to AMA1-C1 7909 in a saline buffer are not inferior to the immune responses to AMA-C1 + CPG 7909 in a phosphate buffer.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Johns Hopkins University Bloomberg School of Public Health, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Narum DL, Thomas AW. Differential localization of full-length and processed forms of PF83/AMA-1 an apical membrane antigen of Plasmodium falciparum merozoites. Mol Biochem Parasitol. 1994 Sep;67(1):59-68. doi: 10.1016/0166-6851(94)90096-5. PMID 7838184
- [Background] Crewther PE, Culvenor JG, Silva A, Cooper JA, Anders RF. Plasmodium falciparum: two antigens of similar size are located in different compartments of the rhoptry. Exp Parasitol. 1990 Feb;70(2):193-206. doi: 10.1016/0014-4894(90)90100-q. PMID 2404781
- [Background] Waters AP, Thomas AW, Deans JA, Mitchell GH, Hudson DE, Miller LH, McCutchan TF, Cohen S. A merozoite receptor protein from Plasmodium knowlesi is highly conserved and distributed throughout Plasmodium. J Biol Chem. 1990 Oct 15;265(29):17974-9. PMID 2211675